CLINICAL TRIAL: NCT06817694
Title: Cognitive Behavioral Therapy for Fear of Cancer Recurrence in Women With BRCA1/2 Gene
Acronym: CBT-FCRBRCA1/2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Josée Savard, Researcher, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-7302
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer Susceptibility Gene (BRCA1) Mutation; BRCA2 Mutation; Fear of Cancer Recurrence
Keywords: BRCA1 Mutation; BRCA 2 Mutation; Fear of cancer recurrence; Cognitive-Behavioral Therapy; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention (Experimental): This group will start as soon as 8 persons have been recruited and randomized into the immediate intervention group.
  Interventions: Behavioral: Cognitive-behavioral group therapy
- Waiting list group (Active Comparator): This group will wait for 4 weeks after being recruited before starting the same intervention as the immediate intervention group.
  Interventions: Behavioral: Cognitive-behavioral group therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral group therapy — The intervention consists of a 4-week cognitive-behavioral group therapy. Each session is given online and will last 90-minutes. The intervention has been adapted to the population of women with a cancer and a BRCA1/2 mutation from a behavioral-cognitive therapy for fear of cancer recurrence that already exists and has already been proven effective.

SUMMARY:
The goal of this clinical trial is to determine whether an adapted version of a current cognitive-behavioural group therapy (CBT) protocol for cancer survivors to the specific needs of women who are carriers of the BRCA1/2 genetic mutation will reduce their levels of fear of cancer recurrence. The main questions this study aims to answer are:

* Will the women who have received the adapted CBT be satisfied with it?
* Will there be a significant difference in the women's fear of cancer recurrence and other variables (e.g., depression, anxiety, insomnia, fatigue, quality of life) between the comparison groups?
* Will the effects of the adapted CBT hold over time?
* What are the roles of different etiological mediating variables in the relationship between fear of cancer recurrence and the effects of the adapted CBT on the severity of fear of cancer recurrence?

Researchers will compare the effects of the adapted CBT between the immediate condition and the waitlist condition.

Participants will be:

* Either placed in the immediate condition or the waitlist condition (the participants in the waitlist condition will begin their therapy once the immediate group is done with theirs).
* Taking part in a group CBT session online once a week for four weeks.
* Completing questionnaires pre-intervention, post-intervention, 3 months post-intervention, and 6 months post-intervention.

DETAILED DESCRIPTION:
Research Problem:

Fear of cancer recurrence (FCR) is defined as fear, worry or concern about the possibility that cancer may recur or progress. FCR is among the top three least-satisfied needs of cancer patients. Almost all patients will experience FCR at some point in their care trajectory. While many will experience occasional and easily managed FCR, mainly at the time of medical testing, others will experience severe and persistent FCR if no intervention is offered. However, it is only in the last two decades that researchers have begun to study FCR in greater depth. Although there is no universally accepted definition and criteria yet, it has been estimated that 45% to 55% of patients have clinical or moderate/severe levels of FCR. Furthermore, longitudinal studies have shown that FCR tends to remain stable over time, particularly among those with clinical levels. FCR is associated with psychological disorders such as anxiety and depression, and reduced quality of life. People experiencing FCR are also more likely to consult healthcare professionals and to use psychotropic drugs such as anxiolytics and antidepressants.

Given the high prevalence and persistence of FCR and its possible consequences, it seems essential, from both an individual and societal point of view, to offer effective psychological interventions to patients with high FCR. Several programs have been developed and tested, with promising results. To our knowledge, our program is the only one internationally to have been implemented in routine oncology care. This program is a group cognitive-behavioral therapy (CBT) of 4 sessions of about 2 hours, whose efficacy has been confirmed in an uncontrolled study (pre- vs. post-treatment). Our treatment protocol and materials, combining therapist and participant manuals, have recently been published in English. The program is integrated into routine cancer care at two hospitals of the Quebec region.

A subpopulation of cancer patients that has been overlooked in the FCR literature is those at high risk of recurrence due to a genetic mutation. BRCA1/2 mutation carriers have a much higher risk of developing breast and ovarian cancer, and at a younger age. They also have a greater risk of cancer recurrence (or a second cancer). Women with a BRCA1/2 mutation are particularly vulnerable to high and persistent levels of FCR, that prophylactic surgery is by no means sufficient to eliminate FCR, and that a cost-effective psychological intervention specifically targeting FCR should ideally be offered as a complement to current practices and counseling offered to these patients. A qualitative study confirmed that FCR is a significant problem in these women and that they emphasized the need to develop and provide access to FCR interventions tailored to the needs of BRCA1/2 mutation carriers. Among other things, they mentioned their particular needs in relation to their younger age and greater risk of cancer recurrence, and raised several issues specific to them, such as having to decide whether to give birth to a child, as pregnancy can increase the risk of recurrence for these women, and the fear of leaving their children motherless should the cancer recur. As for the type of support they would need, they spontaneously mentioned the relevance of group sessions to enable them to share their personal experiences with other women going through the same difficulties. This suggests that a group psychotherapy targeting FCR, adapted to the needs of this specific population, should be developed and tested.

Method:

The adaptation of the treatment manual will be carried out iteratively, using a Delphi method and a series of recorded meetings. As a first step, committee members will be asked to familiarize themselves on an individual basis with the content of a number of existing treatment manuals, including that of Savard et al. (2022), and with the results of the qualitative study by Savard et al. (submitted for publication) conducted among women treated for breast cancer and carrying a BRCA1/2 genetic mutation. An initial meeting will be held to pool the adaptation ideas that each member will have gained from reading the documents. Then, the research team will list all the possible modifications identified, and compile a questionnaire evaluating the importance and relevance of each possible adaptation on a Likert-type scale ranging from "0" (not at all) to "5" (extremely relevant/important), with open-ended comments on each. The questionnaire will be administered to a total of 15 clinicians and researchers in psycho-oncology and hereditary cancer. The research team will compile the data obtained and present it to the same panel of experts at a second meeting in the form of graphs (i.e., percentage endorsement of each answer choice) and lists (for open-ended comments).The expert committee will make a selection in order to eliminate or modify the adaptations least well endorsed and those generating the most questions. The research team will compile a second version of the questionnaire with the possible additions retained. It will be administered to the same 15 clinicians and researchers to assess the relevance/importance of each remaining modification option. If necessary, a third round of evaluation using the same procedure will be carried out. The research team will be responsible for making adaptations to both the Therapist's Manual and the Participant's Manual. These will be resubmitted to the expert committee for comment and final approval. If necessary, an additional meeting will be held.

Participants will be recruited by referral from healthcare professionals working in oncology and oncogenetics, and through advertisements placed in various media across Quebec (posters in waiting rooms, flyers, social media, etc.). Women interested in participating in the study should contact the study coordinator by e-mail or telephone. This will be followed by a telephone interview to assess the main eligibility criteria. The eligible participants will be asked to complete the consent form.

A randomization list will be generated by a statistician blind to the study's objectives, hypotheses and procedures. A series of sealed, opaque envelopes containing the results of the randomization will be prepared by an assistant who is also blind to the same aspects of the study. Once the required number of eligible participants to form a group (n = 8) has been reached, the group will be randomized to : 1) immediate CBT-FCR-BRCA1/2; or 2) waiting list condition on a 1:1 ratio. The envelopes will be opened sequentially by the study coordinator, who will contact each participant by telephone to inform them of the group to which they have been assigned and explain the procedure for the next steps according to group.

Participants assigned to the immediate CBT-FCR-BRCA1/2 group will receive 4 weekly group intervention sessions, while those assigned to the control condition will wait for 4 weeks and complete the same battery of questionnaires (post-attendance measurement) again before receiving the intervention in turn. The sessions will last 90-120 min each and will be led by two facilitators, one of whom will be a psychologist specialized in oncology. To increase the feasibility of the project, facilitate the participation of women who are often young, mothers of young children and on the job market, and to be able to offer the intervention to women with a BRCA1/2 genetic mutation from all over Quebec, the sessions will be offered by videoconference (e.g. Zoom). Patients will receive the Participant's Manual (PDF version sent by e-mail or paper version sent by mail) and instructions to read the relevant module after each session. The psychologist chosen to administer the intervention has already received training in CBT for general FCR and is already offering it in her current practice. She will be assisted by another psychologist or intern/trainee in psycho-oncology. For the purposes of this project, both practitioners will receive one-day training on the medical and psychological aspects of hereditary cancers and on adaptations to the FCR treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* 1) Have completed primary treatment for breast or ovarian cancer (with the exception of adjuvant hormone therapy) for at least 3 months but no more than 10 years.
* 2) Be known to carry a BRCA1/2 genetic mutation.
* 3) Have a clinical level of fear of cancer recurrence as defined by a score of 13 or more on the Fear of Cancer Recurrence Inventory severity subscale.
* 4) Be at least 18 years of age.
* 5) be able to read, understand and express herself in French.

Exclusion Criteria:

* 1) Have distant metastases.
* 2) Have a known cognitive disorder.
* 3) Have a known severe psychological disorder (e.g., psychotic disorder, bipolar disorder, substance abuse or dependence disorder).
* 4) Women taking psychotropic medication are eligible, but only if the dosage has been stable for at least one month.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Fear of cancer recurrence inventory (FCRI) | At recruitment, 4 weeks after recruitment, 3 and 6 months post intervention
  The questionnaire includes 38 questions and assess seven aspects associated with fear of cancer recurrence: Triggers, Severity, Psychological Distress, Functioning impairments, Insight, Reassurance and Coping Strategies. Total values vary between 0 and 152. Higher scores indicate a greater fear of recurrence.

SECONDARY OUTCOMES:
Hospital anxiety and depression scale | At recruitment, 4 weeks after recruitment, 3 and 6 months post intervention
  Includes a total of 14 questions: 7 for anxiety and 7 for depression. For both aspects, the maximum score possible is 21. A score between 0 and 7 indicates a normal level of symptoms, a score between 8 and 10 indicates a borderline abnormal level of symptoms and a score between 11 and 21 indicates an abnormal level of symptoms.
Insomnia severity index (ISI) | At recruitment, 4 weeks after recruitment, 3 and 6 months post intervention
  Includes a total of 7 items. Total score varies between 0 and 28. A score between 0 and 7 indicates no clinically significant insomnia, a score between 8 and 14 indicates subthreshold insomnia, a score between 15 and 21 indicates moderate insomnia (moderate severity) and a score between 22 and 28 indicates clinical insomnia (severe).
Fatigue symptom inventory (FSI) | At recruitment, 4 weeks after recruitment, 3 and 6 months post intervention
  Includes a total of 7 items. Total score varies between 0 and 70. Lower scores indicate lower levels of fatigue and higher scores indicate higher levels of fatigue.
European Organisation for Research and Treatment of cancer's quality of life questionnaire (QLQ-C30) | At recruitment, 4 weeks after recruitment, 3 and 6 months post intervention
  30-items questionnaire developed to assess the quality of life of all cancer patients. Scores range from 0 to 100. A higher score represents a higher level of functioning or a higher level of symptoms, depending on the items.
Revised Illness Perception Questionnaire | At recruitment, 4 weeks after recruitment, 3 and 6 months post intervention
  8 subsections. No total score.
  1. Identity. Score between 0 and 14. Higher score indicates a higher number of symptoms.
  2. Timeline. Higher score = strongly held negative beliefs about the chronicity of the illness.
  3. Consequences. Higher score = strongly held beliefs about the negative consequences of the illness.
  4. Personal control. Higher score = positive beliefs about the controllability of the illness.
  5. Treatment control. Higher score = positive beliefs about the effectiveness of treatment to improve the illness and/or to control the symptoms.
  6. Coherence. Higher score = positive beliefs about the personal understanding of the illness.
  7. Cyclical timeline. Score between 4 and 20. Higher score = strong negative beliefs about the cyclical nature of the illness.
  8. Emotional representation. A higher score = more negative emotions related to the illness.
  Score between 5 and 25 for subscale 2, 5, 6. Score between 6 and 30 for subscale 3, 4, 8.
Intolerance of Uncertainty Scale | At recruitment, 4 weeks after recruitment, 3 and 6 months post intervention
  27-item questionnaire rated on a 5-point Likert scale ranging from 1 (not at all characteristic of me) to 5 (entirely characteristic of me). Total score is obtained by adding up the responses of the items. Total score may vary from 27 to 135. The higher the score, the higher the severity level of intolerance to uncertainty.
Pourquoi s'inquiéter face à la santé (French questionnaire that is not translated in english) | At recruitment, 4 weeks after recruitment, 3 and 6 months post intervention
  25-item questionnaire developed to assess the beliefs related to the worries about the illness. Items are divided in 5 subscales, subscale scores varying between 5 and 25 and each subscale assessing why a person might worry. Higher scores indicate reasons why a person worries.
The Cognitive Avoidance Questionnaire | At recruitment, 4 weeks after recruitment, 3 and 6 months post intervention
  25-item questionnaire rated on a 5-point Likert scale ranging from 1 (not at all corresponding) to 5 (entirely corresponding). Total score varies between 25 and 125. The higher the score, the higher the level of cognitive avoidance.
Worry Behaviors Inventory | At recruitment, 4 weeks after recruitment, 3 and 6 months post intervention
  10-item questionnaire rated with a Likert-like scale ranging from 0 (none of the time) to 4 (all of the time). Total scores vary from 0 to 40, a higher score indicating a higher level of worry behaviors.
Reassurance Seeking Behaviour subscale in the Health Anxiety Questionnaire | At recruitment, 4 weeks after recruitment, 3 and 6 months post intervention
  3-item subscale with a Likert-like subscale ranging from 0 (not at all or rarely) to 3 (most of the time). Total score varies from 0 to 9, a higher score indicating a higher need for reassurance seeking behaviors.
Reassurance Questionnaire | At recruitment, 4 weeks after recruitment, 3 and 6 months post intervention
  10-item questionnaire assessing the extent to which patients report feeling reassured by their attending physician. Questions are rated from not at all to most of the time. Scores vary from 10 to 40. The higher the score, the lower the feeling of reassurance.
Importance of Staying in Control Subscale of the Beliefs About Losing Control Inventory | At recruitment, 4 weeks after recruitment, 3 and 6 months post intervention
  3-item subscale rated with a Likert-like scale ranging from 0 (not at all) to 4 (very much). Total score varies between 0 and 12. A higher score indicates a greater importance given to staying in control.

REFERENCES:
- [Background] Lebel S, Ozakinci G, Humphris G, Mutsaers B, Thewes B, Prins J, Dinkel A, Butow P; University of Ottawa Fear of Cancer Recurrence Colloquium attendees. From normal response to clinical problem: definition and clinical features of fear of cancer recurrence. Support Care Cancer. 2016 Aug;24(8):3265-8. doi: 10.1007/s00520-016-3272-5. Epub 2016 May 12. PMID 27169703
- [Background] Simard S, Thewes B, Humphris G, Dixon M, Hayden C, Mireskandari S, Ozakinci G. Fear of cancer recurrence in adult cancer survivors: a systematic review of quantitative studies. J Cancer Surviv. 2013 Sep;7(3):300-22. doi: 10.1007/s11764-013-0272-z. Epub 2013 Mar 10. PMID 23475398
- [Background] Baker F, Denniston M, Smith T, West MM. Adult cancer survivors: how are they faring? Cancer. 2005 Dec 1;104(11 Suppl):2565-76. doi: 10.1002/cncr.21488. PMID 16258929
- [Background] Armes J, Crowe M, Colbourne L, Morgan H, Murrells T, Oakley C, Palmer N, Ream E, Young A, Richardson A. Patients' supportive care needs beyond the end of cancer treatment: a prospective, longitudinal survey. J Clin Oncol. 2009 Dec 20;27(36):6172-9. doi: 10.1200/JCO.2009.22.5151. Epub 2009 Nov 2. PMID 19884548
- [Background] Savard J, Ivers H. The evolution of fear of cancer recurrence during the cancer care trajectory and its relationship with cancer characteristics. J Psychosom Res. 2013 Apr;74(4):354-60. doi: 10.1016/j.jpsychores.2012.12.013. Epub 2013 Jan 26. PMID 23497839
- [Background] Savard J, Filion C, Brearty CM, Caplette-Gingras A, Chiquette J, Dorval M. Fear of cancer recurrence in breast cancer survivors carrying a BRCA1/2 mutation: A qualitative study. Cancer Med. 2024 Jan;13(1):e6889. doi: 10.1002/cam4.6889. Epub 2024 Jan 8. PMID 38192174
- [Background] Champagne A, Ivers H, Savard J. Utilization of health care services in cancer patients with elevated fear of cancer recurrence. Psychooncology. 2018 Aug;27(8):1958-1964. doi: 10.1002/pon.4748. Epub 2018 Jun 1. PMID 29719072
- [Background] Butow PN, Turner J, Gilchrist J, Sharpe L, Smith AB, Fardell JE, Tesson S, O'Connell R, Girgis A, Gebski VJ, Asher R, Mihalopoulos C, Bell ML, Zola KG, Beith J, Thewes B. Randomized Trial of ConquerFear: A Novel, Theoretically Based Psychosocial Intervention for Fear of Cancer Recurrence. J Clin Oncol. 2017 Dec 20;35(36):4066-4077. doi: 10.1200/JCO.2017.73.1257. Epub 2017 Nov 2. PMID 29095681
- [Background] Lebel S, Maheu C, Lefebvre M, Secord S, Courbasson C, Singh M, Jolicoeur L, Benea A, Harris C, Fung MF, Rosberger Z, Catton P. Addressing fear of cancer recurrence among women with cancer: a feasibility and preliminary outcome study. J Cancer Surviv. 2014 Sep;8(3):485-96. doi: 10.1007/s11764-014-0357-3. Epub 2014 Apr 23. PMID 24756313
- [Background] Smith AB, Costa D, Galica J, Lebel S, Tauber N, van Helmondt SJ, Zachariae R. Spotlight on the Fear of Cancer Recurrence Inventory (FCRI). Psychol Res Behav Manag. 2020 Dec 21;13:1257-1268. doi: 10.2147/PRBM.S231577. eCollection 2020. PMID 33376421
- [Background] Savard, J., Caplette-Gingras, A., Casault, L., & Hains, J. Treating Fear of Cancer Recurrence with Group Cognitive-behavioral Therapy: A Step-by-step Guide: Springer; 2022.
- See also: Humphris, G., & Rogers, S. (2012). AFTER and beyond: cancer recurrence fears and a test of an intervention in oral and oropharyngeal patients. Social Science and Dentistry, 2(1), 29-38. — https://ssdopen.com/media/articles/AFTER_and_beyond__cancer_recurrence_fears_and_a_test_of_an_intervention_in_oral_and_oropharyngeal_patients.pdf
- See also: Savard, J., Savard, M.-H., Caplette-Gingras, A., Casault, L., & Camateros, C. (2018). Development and feasibility of a group cognitive-behavioral therapy for fear of cancer recurrence. Cognitive and Behavioral Practice, 25(2), 275-285. — https://doi.org/https://doi.org/10.1016/j.cbpra.2017.08.001